CLINICAL TRIAL: NCT04877613
Title: Phase I Trial of GFRα4 CAR T Cells in Adult Patients With Recurrent or Metastatic Medullary Thyroid Cancer
Brief Title: GFRα4 CAR T Cells in MTC Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB# 848848; UPCC# 12320
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Medullary Thyroid Cancer; Recurrent Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: The is a Phase I dose finding study to determine the safety of CART-GFRa4 cells. Dose escalation and determination of maximum tolerated dose (MTD) will be based on the standard 3+3 design to explore 3 possible dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: single dose of 5x10^7 CART-GFRa4 cells via intravenous infusion (Experimental)
  Interventions: Drug: single dose of CART-GFRa4 cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Cohort -1: single dose of 2x10^7 CART-GFRa4 cells via intravenous infusion (Experimental)
  Interventions: Drug: single dose of CART-GFRa4 cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Cohort 2: single dose of 1x10^8 CART-GFRa4 cells via intravenous infusion (Experimental)
  Interventions: Drug: single dose of CART-GFRa4 cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Cohort 3: single fixed dose of 3x10^8 CART-GFRa4 cells via intravenous infusion (Experimental)
  Interventions: Drug: single dose of CART-GFRa4 cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: single dose of CART-GFRa4 cells — Intravenous infusion of lentiviral transduced autologous T cells that have been engineered to express an extracellular single chain antibody (scFv) with specificity towards GFRa4 with fludarabine and cyclophosphamide.
Drug: Fludarabine — Lymphodepletion
Drug: Cyclophosphamide — Lymphodepletion

SUMMARY:
This is an open-label phase 1 study to assess the safety and feasibility of autologous T cells expressing a single-chain scFv targeting GFRα4 with tandem TCR/CD3ζ and 4-1BB (TCRζ/4-1BB) co-stimulatory domains (referred to as "CART-GFRa4 cells") in patients with incurable medullary thyroid cancer (MTC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent
2. Male or female age ≥ 18 years
3. Histologically or cytologically confirmed diagnosis of medullary thyroid cancer (MTC).
4. Incurable recurrent/metastatic disease that is progressive after at least 1 prior tyrosine kinase inhibitor (TKI) containing regimen, or the patient was intolerant of or declined such therapy.
5. Adequate organ function defined as:

   1. Serum creatinine ≤ 2.5 mg/dl or estimated creatinine clearance ≥ 30 ml/min and not on dialysis.
   2. AST ≤ 5x upper limit of normal range and total bilirubin ≤ 2.0 mg/dl; except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome.
   3. Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO/MUGA
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen greater than 92% on room air.
6. ECOG Performance Status that is either 0 or 1.
7. Toxicities from prior therapies must have recovered to grade ≤ 2 according to the CTCAE 5.0 criteria or to the patient's prior baseline.
8. Patients must have evaluable disease as defined by RECIST 1.1.
9. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Evidence of active hepatitis B or hepatitis C infection. The following would not qualify as an active infection, thus would not exclude the subject from participating

   1. Positive HBV serology with undetectable viral load and ongoing antiviral prophylaxis for potential HBV reactivation.
   2. Positive HCV serology with quantitative PCR for plasma HCV RNA below the lower limit of detection, with or without concurrent antiviral HCV treatment.
2. Any other active, uncontrolled infection.
3. Any prior history of moderate to severe (Grade 2 or higher) pneumonitis.
4. Subjects with chronic kidney disease with Grade 2 or higher renal impairment (eGFR or CrCl 59-30 ml/min/1.73 m2).
5. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
6. Clinically apparent arrhythmia or arrhythmias that are not stable on medical management within two weeks of physician-investigator confirmation of eligibility.
7. Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (≤10mg equivalent of prednisone). Use of inhaled steroids is allowable. Corticosteroid treatment as anti-emetic prophylaxis on the day of lymphodepleting chemotherapy administration is allowed per institutional practice.
8. Any moderate to severe skin rash or allergies requiring systemic treatment.
9. Receipt of immune checkpoint inhibitors within 2 months prior to physician-investigator confirmation of eligibility - Retired with Protocol Version 3.
10. Pregnant or nursing (lactating) women.
11. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg daily of prednisone. Patients with autoimmune neurological diseases (such as MS or Parkinson's) will be excluded.
12. Have any history of prior or active central nervous system (CNS) involvement (e.g., leptomeningeal disease, parenchymal masses) with MTC. Screening for this (e.g., with lumbar puncture and/or brain MRI) is not required unless suspicious symptoms and/or radiographic findings are present. Subjects with calvarial metastatic disease that extends intracranially and involves the dura will be excluded, even if CSF is negative for MTC.
13. Known seizure disorder or history of prior seizures requiring medication.
14. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2039-06-01 (Estimated); Study Completion 2039-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0. | 15 years

SECONDARY OUTCOMES:
Percentage of manufacturing products that meet release criteria. | 3 months
Number of subjects who have a response (ORR) | 12 months
Best Overall Response (BOR) | 12 months
Duration of Response (DOR) | 12 months
Overall survival (OS) | 12 months
Progression-free survival (PFS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Cohen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No